CLINICAL TRIAL: NCT00914849
Title: A Phase II Study Evaluating the Safety and Efficacy of Intravenous AMD3100 for the Mobilization and Transplantation of HLA-Matched Sibling Donor Hematopoietic Stem Cells in Patients With Advanced Hematological Malignancies
Brief Title: Intravenous (IV) AMD3100 for Mobilization and Matched Related Transplant for Advanced Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0713 / 201103429
Record Dates: First submitted 2009-06-01; First posted 2009-06-05 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms | interventions — plerixafor; Leukapheresis; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - Donor (Experimental): * Day 1
    * AMD3100 320 ug/kg IV
    * Leukopheresis
  * Day 2 (if peripheral blood stem cell (PBSC) collected is not sufficient)
    * AMD3100 320 ug/kg IV
    * Leukopheresis
  Interventions: Drug: AMD3100; Procedure: Leukopheresis
- Arm 2 - Recipient (Experimental): Standard of care and physician choice myeloablative or non-myeloablative chemotherapy with or without total body irradiation (permitted = cyclophosphamide and single dose total body irradiation (TBI) / fludarabine and busulfan / fractionated TBI and cyclophosphamide / fractionated TBI, etoposide, and cyclophosphamide / busulfan and cyclophosphamide / fludarabine, busulfan, and ATGAM
  Day 0 = Stem Cell Transplant
  Interventions: Procedure: Stem cell transplant

INTERVENTIONS:
Drug: AMD3100
  Other Names: Mozobil; Plerixafor
  Arms: Arm 1 - Donor
Procedure: Leukopheresis
  Arms: Arm 1 - Donor
Procedure: Stem cell transplant
  Arms: Arm 2 - Recipient

SUMMARY:
To reduce the number of donors treated with IV AMD3100 who require a second collection to obtain the minimum cells necessary for allogeneic stem cell transplant.

DETAILED DESCRIPTION:
* To reduce the number of donors treated with intravenous (IV) AMD3100 who require a second collection to obtain the minimum CD34/kg (2 X 106) necessary for allogeneic stem cell transplantation when compared to our historic group who received 240ug SC AMD3100 from 33% (8 in 24) to 11% (3 in 27).
* To estimate with 95% confidence intervals the proportion of human leukocyte antigen (HLA)-identical sibling donors who experience grade 3-4 infusional toxicity and the proportion from whom ≥ 2.0 x 10e6 CD34+ cells/kg recipient weight are safely mobilized following one or two intravenous infusions.
* To determine the kinetics of stem cell and lymphocyte mobilization using IV AMD3100 and to determine if peripheral blood stem cell products collected after mobilization with IV AMD3100 can be used safely for hematopoietic cell transplantation in HLA-matched recipients as measured by neutrophil engraftment by day +21.
* To determine the pharmacokinetics and pharmacodynamics of IV AMD3100 on stem cell and T-cell phenotyping and on immune reconstitution after transplantation.
* To determine the rate of acute graft-versus-host disease (GVHD) and chronic GVHD in patients who receive IV AMD3100 mobilized peripheral blood stem cells.

ELIGIBILITY:
Inclusion Criteria:

Donor Eligibility

* Donor is 18 to 70 years of age inclusive.
* If female and of child-bearing age: must be non-pregnant, not breast feeding and agree to use adequate contraception.
* Donor is a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Donor must be willing to provide written informed consent.
* Adequate cardiac function with no history of congestive heart failure and no history of atrial fibrillation or ventricular tachyarrhythmia.
* Adequate renal function as defined by a calculated serum creatinine clearance of ≥75% of normal (Cockcroft-Gault equation).
* Adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis.
* Adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality. No history of cerebrovascular accident or seizure disorder requiring anticonvulsant medication.
* Donor must be HIV-1&2 antibody and HTLV-I&II antibody sero-negative, by Food and Drug Administration (FDA) licensed test.
* Donor must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Donor must demonstrate ability to be compliant with study regimen.
* Donor must not have an active infection at the time of study entry.
* Donor does not have active alcohol or substance abuse within 6 months of study entry.
* Donor is not currently enrolled on another investigational agent study.
* Donor does not have any medical condition, which, in the opinion of the clinical investigator, would interfere with his/her evaluation.

Recipient Eligibility

* Recipient must have available the successful collection of an AMD3100 mobilized product. When an adequate collection cannot be obtained using G-CSF, some recipients may need to receive a combined product of mobilized cells with AMD3100 and g granulocyte-colony stimulating factor (G-CSF). Recipients who receive less than 2.0 X 106 CD34+ cells/kg/actual recipient weight after two days of IV AMD3100 will not be considered "eligible" but followed per protocol for safety purposes only.
* Patient is 18 to 65 years of age inclusive.
* Patient is willing and has a 6/6 HLA-matched sibling willing to donate PBSC for transplant.
* Patient must provide signed informed consent.
* If female and of child-bearing age: must be non-pregnant, not breast feeding, and uses adequate contraception.
* Patient must have one of the following diagnoses:

  * Acute myelogenous leukemia (AML) in 1st or subsequent remission or in relapse,
  * Acute lymphoblastic leukemia (ALL) in 1st or subsequent remission or in relapse,
  * Myelodysplastic syndrome either intermediate 1 or 2, or high risk by the International Prognostic Scoring System,
  * Chronic myelogenous leukemia (CML) in accelerated or second chronic phase,
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission, or refractory relapse,
  * Chronic lymphocytic leukemia (CLL), Rai Stage 2-4, failing at least 2 prior regimens, OR
  * Multiple myeloma (MM), Stage 2-3.
* Adequate cardiac function with a left ventricular ejection fraction ≥ 40%.
* Adequate pulmonary function defined as NO severe or symptomatic restrictive or obstructive lung disease, and formal pulmonary function testing showing an FEV1 ≥50% of predicted and a DLCO ≥40% of predicted, corrected for hemoglobin.
* Adequate renal function as defined by a serum creatinine clearance of ≥75% of normal (Cockcroft-Gault equation).
* Adequate hepatic function as defined by a total bilirubin <2x normal or absence of hepatic fibrosis/cirrhosis.
* Adequate neurologic function as defined by NO evidence of a severe central or peripheral neurologic abnormality. Patients with a history of previous central nervous system (CNS) tumor involvement are eligible provided they are without symptoms or signs and the CNS is now free of disease on lumbar puncture and CT scan of the brain.
* No evidence of active infection at the time of the transplant preparative regimen or at time of transplantation.
* Patient must be HIV-1&2 antibody and HTLV-I & II antibody sero-negative, by FDA licensed test.
* Patient has an ECOG performance status of 0 or 1.
* Patient must demonstrate ability to be compliant with medical regimen.
* Patient must not have active alcohol or substance abuse within 6 months of study entry.
* Patient must not be enrolled on another investigational agent concurrently.
* Patient must not have any medical condition, which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient.

Exclusion Criteria:

* See Inclusion criteria above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John DiPersio, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levesque JP, Hendy J, Takamatsu Y, Simmons PJ, Bendall LJ. Disruption of the CXCR4/CXCL12 chemotactic interaction during hematopoietic stem cell mobilization induced by GCSF or cyclophosphamide. J Clin Invest. 2003 Jan;111(2):187-96. doi: 10.1172/JCI15994. PMID 12531874
- [Background] Peled A, Petit I, Kollet O, Magid M, Ponomaryov T, Byk T, Nagler A, Ben-Hur H, Many A, Shultz L, Lider O, Alon R, Zipori D, Lapidot T. Dependence of human stem cell engraftment and repopulation of NOD/SCID mice on CXCR4. Science. 1999 Feb 5;283(5403):845-8. doi: 10.1126/science.283.5403.845. PMID 9933168
- [Background] Broxmeyer HE, Hangoc G, Cooper S, Bridger G. Interference of the SDF-1/CXCR4 axis in mice with AMD3100 induces rapid high level mobilization of hematopoietic progenitor cells, and AMD3100 acts synergistically with G-CSF and MIP-1 alpha to mobilize progenitors. Blood. 2001;96:3371a
- [Background] Broxmeyer HE, Hangoc G, Cooper S, Li X, Bridger G, Clapp DW. AMD3100, an antagonist of CXCR4 and mobilizer of myeloid progenitor cells, is a potent mobilizer of competitive repopulating long term marrow self renewing stem cells in mice. Blood. 2002;98:2397a
- [Background] Liles WC, Broxmeyer HE, Rodger E, Wood B, Hubel K, Cooper S, Hangoc G, Bridger GJ, Henson GW, Calandra G, Dale DC. Mobilization of hematopoietic progenitor cells in healthy volunteers by AMD3100, a CXCR4 antagonist. Blood. 2003 Oct 15;102(8):2728-30. doi: 10.1182/blood-2003-02-0663. Epub 2003 Jul 10. PMID 12855591
- [Background] Devine S, Adkins D, Khoury H, Vij R, Goodnough LT, Graubert T, Tomasson M, Blum W, DiPersio J, Brown R. Mobilization of donors with GM-CSF plus G-CSF or GM-CSF alone results in significantly different graft composition compared to G-CSF alone. Blood. 2002;100:825a
- [Background] Devine SM, Vij R, Rettig M, Todt L, McGlauchlen K, Fisher N, Devine H, Link DC, Calandra G, Bridger G, Westervelt P, Dipersio JF. Rapid mobilization of functional donor hematopoietic cells without G-CSF using AMD3100, an antagonist of the CXCR4/SDF-1 interaction. Blood. 2008 Aug 15;112(4):990-8. doi: 10.1182/blood-2007-12-130179. Epub 2008 Apr 21. PMID 18426988
- [Background] Broxmeyer HE, Orschell CM, Clapp DW, Hangoc G, Cooper S, Plett PA, Liles WC, Li X, Graham-Evans B, Campbell TB, Calandra G, Bridger G, Dale DC, Srour EF. Rapid mobilization of murine and human hematopoietic stem and progenitor cells with AMD3100, a CXCR4 antagonist. J Exp Med. 2005 Apr 18;201(8):1307-18. doi: 10.1084/jem.20041385. PMID 15837815
- [Background] Hess DA, Bonde J, Craft TP, Wirthlin L, Hohm S, Lahey R, Todt LM, Dipersio JF, Devine SM, Nolta JA. Human progenitor cells rapidly mobilized by AMD3100 repopulate NOD/SCID mice with increased frequency in comparison to cells from the same donor mobilized by granulocyte colony stimulating factor. Biol Blood Marrow Transplant. 2007 Apr;13(4):398-411. doi: 10.1016/j.bbmt.2006.12.445. PMID 17382247
- [Derived] Schroeder MA, Rettig MP, Lopez S, Christ S, Fiala M, Eades W, Mir FA, Shao J, McFarland K, Trinkaus K, Shannon W, Deych E, Yu J, Vij R, Stockerl-Goldstein K, Cashen AF, Uy GL, Abboud CN, Westervelt P, DiPersio JF. Mobilization of allogeneic peripheral blood stem cell donors with intravenous plerixafor mobilizes a unique graft. Blood. 2017 May 11;129(19):2680-2692. doi: 10.1182/blood-2016-09-739722. Epub 2017 Mar 14. PMID 28292947
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 08/12/2009 and closed to participants enrollment on 01/31/2011.
Groups:
- Arm 1 - Donor: * Day 1
    * AMD3100 320 ug/kg intravenous (IV)
    * Leukopheresis
  * Day 2 (if peripheral blood stem cell (PBSC) collected is not sufficient)
    * AMD3100 320 ug/kg IV
    * Leukopheresis
Period: Overall Study
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Started | 34 | 34
Completed | 33 | 33
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not eligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: One recipient was not transplanted because of donor withdrawal of consent to collect a second day after a failed first day apheresis attempt.
Groups:
- Arm 1 - Donor: * Day 1
    * AMD3100 320 ug/kg IV
    * Leukopheresis
  * Day 2 (if PBSC collected is not sufficient)
    * AMD3100 320 ug/kg IV
    * Leukopheresis
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Median (Full Range); unit: years] | 50 [28 to 65] | 54 [25 to 68] | 52 [25 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Donors Treated With IV AMD3100 Who Required a Second Collection to Obtain the Minimum CD34/kg (2 X 106) Necessary for Allogeneic Stem Cell Transplant
Time Frame: Completion of enrollment of all donors (17 months)
Population: 3 donors failed to reach target after two collections and 1 donor withdrew consent after failing to reach the goal on the first collection.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 29 | 0
participants | 10 |

2. Secondary Outcome: Number of Donors Who Experience Grade 3-4 Infusional Toxicity
Time Frame: Up to Day 2
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 34 | 0
participants | 0 |

3. Secondary Outcome: Number of Recipients Who Have Neutrophil Engraftment
Time Frame: Day 21
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
participants |  | 33

4. Secondary Outcome: Pharmacokinetics of IV AMD3100 as Measured by the Mean Maximum Plasma Concentration (Cmax)
Description: -Blood samples for pharmacokinetics were drawn on the following schedule:
  * prior to IV infusion
  * 15 minutes after start of infusion
  * 30 minutes after start of infusion
  * 1 hour after start of infusion
  * 4 hours after start of infusion
  * 6 hours after start of infusion
  * 9 hours after start of infusion
  * 24 hours after start of infusion
Time Frame: Day 1 and Day 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 34 | 0
ng/mL | 1391 (488) |

5. Secondary Outcome: Pharmacokinetics of IV AMD3100 as Measured by Half Life
Description: as for outcome 4
Time Frame: Day 1 and Day 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 34 | 0
hours | 5.42 (1.24) |

6. Secondary Outcome: Pharmacokinetics of IV AMD3100 as Measured by Mean Area Under Curve (AUC)
Time Frame: Day 1 and Day 2
Measure: Mean (Standard Deviation); unit: hr.ng/mL
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 34 | 0
hr.ng/mL | 5049 (1233) |

7. Secondary Outcome: Rate of Acute GVHD (Grade II-IV) in Recipients
Time Frame: Day 0-Day 100 (acute)
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
participants |  | 4

8. Secondary Outcome: Rate of Acute GVHD (Grade III-IV) in Recipients
Time Frame: Day 0-Day 100 (acute)
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
participants |  | 4

9. Secondary Outcome: Time to Neutrophil Engraftment for Recipients
Description: Measured by determine the first 3 consecutive measurement of neutrophil count = 500/ul following conditioning regimen induced nadir.
Time Frame: Up through Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
days |  | 14 [11 to 24]

10. Secondary Outcome: Time to Platelet Engraftment for Recipients
Description: Measured by determining the first of 3 consecutive measurements of platelet count = 20,000/ul without platelet transfusion support for 7 days.
Time Frame: Up to Day 100
Measure: Median (Full Range); unit: days
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
days |  | 25 [15 to 219]

11. Secondary Outcome: Transplant Related Mortality Rate for Recipients
Description: Death that results from a transplant procedure related complication rather than from relapse of the underlying disease or unrelated cause.
Time Frame: Day 100
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 33
participants |  | 1

12. Secondary Outcome: Grade 3-4 Toxicity for Recipients
Description: Assessed and graded according to NCI Common Terminology for Adverse Events Version 3.0.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 34
participants
  Grade 3 fatigue |  | 3
  Grade 3 thrombocytopenia |  | 1
  Grade 3 mucositis |  | 5
  Grade 3 GI fistula |  | 1
  Grade 3 increased transaminase |  | 2
  Grade 3 febrile neutropenia |  | 32
  Grade 3 bacteremia+ |  | 4
  Grade 3 respiratory distress |  | 1
  Grade 3 renal failure |  | 6

13. Secondary Outcome: Rate of Chronic GVHD in Recipients
Time Frame: Day 101-1 year
Population: 8 patients are not evaluable because they were not alive for the outcome measure time frame.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 0 | 25
participants |  | 7

14. Secondary Outcome: Number of Donors Who Experience Grade 3-4 Mobilization Toxicity Due to Pheresis Procedure
Time Frame: Up to Day 2
Measure: Number; unit: participants
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Number analyzed (Participants) | 34 | 0
participants | 2 |

ADVERSE EVENTS:
Arm/Group | Arm 1 - Donor | Arm 2 - Recipient
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 33/33 | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Donor (N=33) | Arm 2 - Recipient (N=33)
Abdominal cramping (Gastrointestinal disorders) | 17 | 0
Adult respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bacteremia (Infections and infestations) | 0 | 4
Catheter site infection (Infections and infestations) | 0 | 3
Catheter site pain (General disorders) | 0 | 5
Chest pain (Cardiac disorders) | 2 | 0
Cold sensation (General disorders) | 3 | 0
Congestive heart failure (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 12 | 16
Distension/abdominal bloating (Gastrointestinal disorders) | 10 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Fatigue (General disorders) | 0 | 13
Febrile neutropenia (Infections and infestations) | 0 | 32
Fever (General disorders) | 0 | 2
GI fistula (Gastrointestinal disorders) | 0 | 1
Generalized weakness (General disorders) | 0 | 30
Hand tremor (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 7
Hematuria (Renal and urinary disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 2
Hyperbiluribinemia (Investigations) | 0 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 14
Hypertension (Vascular disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 24 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 8
Hypotension (Vascular disorders) | 7 | 3
Incontinence (Renal and urinary disorders) | 0 | 1
Increase transaminase (Investigations) | 0 | 8
Insomnia (Psychiatric disorders) | 4 | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Lightheadedness (Nervous system disorders) | 5 | 0
Lower extremities edema (General disorders) | 0 | 13
Mental status change (Psychiatric disorders) | 0 | 2
Mucositis (Gastrointestinal disorders) | 0 | 18
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Parotiditis (Infections and infestations) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 6
Sensory neuropathy (Nervous system disorders) | 23 | 0
Sinus bradycardia (Cardiac disorders) | 8 | 0
Skin nodules (Skin and subcutaneous tissue disorders) | 0 | 1
Sweating (diaphoresis) (General disorders) | 5 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Thrombocytopenia (Investigations) | 4 | 2
Thrombosis/embolism (DVT) (Vascular disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 3
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Vasovagal episode (Nervous system disorders) | 6 | 0
Vomiting (Gastrointestinal disorders) | 0 | 12
Warm sensation (General disorders) | 1 | 0
Weight loss (Investigations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes